CLINICAL TRIAL: NCT00914420
Title: OCT Evaluation of Stent Struts Re-endothelization in Patients With Acute Coronary Syndromes: a Comparison of the Intrepide™ Stent vs. Taxus™
Brief Title: Optical Coherence Tomography (OCT) Evaluation of Re-endothelization: A Comparison of the Intrepide™ Stent Versus Taxus™
Acronym: OISTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clearstream Technologies Ltd. (Industry)
Responsible Party: Dr Giuseppe Sangiorgi Dr Antonio Colombo, University Hospital Modena - Italy ; Raffaele hospital, Milano- Italy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CST10
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2010-04

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: OCT; Reendothelialisation; Intrepide; Trapidil; Taxus
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrepide (Experimental): Group A- Primary stenting with Intrepide trapidil eluting stent
  Interventions: Device: Intrepide Trapidil eluting stent
- Taxus (Experimental): Group B Stenting with Taxus DES
  Interventions: Device: Taxus drug eluting stent

INTERVENTIONS:
Device: Intrepide Trapidil eluting stent — The INTREPIDE coronary stent system consists of a balloon expandable stent coated with two layers of Trapidil and parylene. The Trapidil eluting stent is pre-mounted on a Nimbus PCTA balloon and is intended for use in the treatment of CAD.
  The controlled release of Trapidil is achieved through the parylene barrier, locally delivering the drug to the target lesion, inhibiting smooth muscle cell proliferation and hence neointimal hyperplasia.
  Arms: Intrepide
Device: Taxus drug eluting stent — Paclitaxel Drug eluting stent manufactured by Boston Scientific
  Arms: Taxus

SUMMARY:
Patients presenting with ACS (Acute Coronary Syndrome) in the emergency department will be screened for clinical eligibility and asked to sign informed consent to the study.

A total of 40 patients will be randomized. 20 of them will receive a Trapidil eluting stent (Intrepide™ stent), 20 will receive a Paclitaxel eluting stent (Taxus™ stent). After 90 days the patients who were treated with the INTREPIDE stent in the first lesion will be treated with the Taxus stent in the second lesion. After 90 days the patients who were treated with the Taxus stent in the first lesion will be treated with the INTREPIDE stent in the second lesion.

Coronary angiography will be performed through the femoral (groin) or radial (wrist) artery with the use of standard techniques. The doctor will determine if the patient is qualified for enrolment at the end of the diagnostic coronary angiogram

ELIGIBILITY:
Inclusion Criteria:

Clinical

* >18 years of age,
* symptoms of non ST-elevation ACS (defined by the ACC/AHA criteria) for 30 min but <48 h
* Patient must provide written informed consent prior to the procedure using a form that is approved by the local Institutional Review Board

Angiographic

* reference vessel diameter of culprit/target lesion between 2.25 to 3.5 mm (visual estimate)
* discrete target lesion (maximum length of 28 mm by visual estimation)
* target lesion is in a native coronary artery
* presence of another lesion more than 70% in a vessel different from the culprit one amenable of planned percutaneous treatment 90 days thereafter.

Exclusion Criteria:

Clinical

* previously documented left ventricular ejection fraction of less than 30%
* estimated life expectancy of less than 12 months
* a history of bleeding diathesis, leukopenia, thrombocytopenia, or severe hepatic or renal dysfunction
* participation in another study
* inability to give informed consent owing to prolonged cardiopulmonary resuscitation
* and dominant Renal impairment (serum creatinine > 2.0 mg/dl) Angiographic
* non-culprit lesion located in the proximal LAD or in a proximal and dominant Circumflex artery
* previous PCI of the target vessels restenosis or stent thrombosis as culprit lesion
* unprotected left main coronary artery disease
* non-culprit lesion located in a vein graft
* severe multivessel disease (three major epicardial vessel disease) need of overlapping stenting for one lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-11 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
To compare stent re-endothelialization using Trapidil drug eluting stent versus Taxus paclitaxel eluting stent at 3 months after intervention. The primary endpoint will be defined by % of stent struts neointimal coverage at 90 days | 3 months

SECONDARY OUTCOMES:
In-stent binary angiographic restenosis and in-stent late lumen loss; in segment late loss; assessed by quantitative computed angiography (QCA) at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Columbo, MD, Principal Investigator — San Raffaele hospital, Milano; Giuseppe M Sangiorgi, MD, Principal Investigator — University Hospital Modena Italy
Locations (1):
- University Hospital Modena, Modena, Italy

REFERENCES:
- See also: Industry Sponsor — http://www.clearstream.ie